CLINICAL TRIAL: NCT00199108
Title: A Phase-2 Clinical Study to Determine the Efficacy and Safety of Depocyt (Cytarabine Liposome Injection) for the Treatment of CNS Relapse in Adult Patients With Acute Lymphoblastic Leukemia or Very Aggressive Lymphoma
Brief Title: Treatment of Acute Lymphoblastic Leukemia or Aggressive Lymphoma With Relapse in Central Nervous System With Depocyt
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Nicola Goekbuget, Principal Investigator, Goethe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMALL06
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Adult Acute Lymphocytic Leukemia
Keywords: CNS relapse; ALL; Treatment
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Dexamethasone

ARMS (1):
- Only 1 arm (Experimental)
  Interventions: Drug: Depocyt; Drug: Dexamethasone

INTERVENTIONS:
Drug: Depocyt
Drug: Dexamethasone

SUMMARY:
Patients with acute lymphoblastic leukaemia or very aggressive lymphoma and documented isolated CNS relapse or CNS relapse combined with other relapse sites should receive therapy with intrathecal DepoCyte at least once. Treatment may be repeated during induction phase each 2 weeks and monthly during maintenance phase. The study aim is to replace the usual 2-3 weekly applications of intrathecal triple therapy with one application of DepoCyte. Primary objective is the response rate after one application of DepoCyte. Further objectives are the compilation of data regarding safety and toxicity

ELIGIBILITY:
Inclusion Criteria:

* proven diagnosis of ALL or very aggressive Non-Hodgkin-Lymphoma (Burkitt/Burkitt-like) and CNS relapse
* CNS involvement demonstrated by a positive ventricular or lumbar CSF cytology or characteristic signs and symptoms of neoplastic meningitis plus an MRI or CT scan indicating the presence of meningeal involvement
* in combined relapse in CNS and other locations: systemic therapy with CNS active drugs can be postponed for at least 2 weeks
* Karnofsky Performance Score is > or = 60%
* 18 years of age or older
* free of uncontrolled infection
* recovered from any grade III / IV toxicities attributable to prior treatment with the exception of hematotoxicity
* patient not pregnant or breast feeding and effective methods to prevent pregnancy
* free from severe heart, lung, liver or kidney dysfunction
* written informed consent

Exclusion Criteria:

* failed to respond (as defined by no clearance of the CSF) to > 1 dose of prior i.th. MTX or ARAC or triple therapy
* history of neurotoxicity (grade III - IV) attributed to i.th. or systemic HD therapy with MTX or ARAC
* prior CNS relapse < 1 month before

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-04 (Actual); Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
response rate after one application of DepoCyte | one cycle

SECONDARY OUTCOMES:
response rate at later time-points, toxicity (WHO), death in induction and CR, time to neurological progression, frequency of improvement in pre-existing meningeal-disease related neurological symptoms, Karnofsky Performance Status, Survival | after each cycle and during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Hoelzer, MD,PhD, Study Chair — University Hospital Frankfurt, Medical Dept. II
Locations (1):
- University Hospital, Medical Dept. II, Frankfurt, Germany

REFERENCES:
- [Background] Gokbuget N, Hartog CM, Bassan R, Derigs HG, Dombret H, Greil R, Hernandez-Rivas JM, Huguet F, Intermesoli T, Jourdan E, Junghanss C, Leimer L, Moreno MJ, Reichle A, Ribera J, Schmid M, Serve H, Stelljes M, Stuhlmann R, Hoelzer D; German Multicenter Study Group for Adult ALL and the European Working Group for Adult ALL. Liposomal cytarabine is effective and tolerable in the treatment of central nervous system relapse of acute lymphoblastic leukemia and very aggressive lymphoma. Haematologica. 2011 Feb;96(2):238-44. doi: 10.3324/haematol.2010.028092. Epub 2010 Oct 15. PMID 20952517